CLINICAL TRIAL: NCT01602835
Title: Human Urine Sample Collection for Alport Nephropathy Biomarker Studies
Status: Terminated | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPLATFRM2201
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Alport Syndrome
Keywords: Alport syndrome; proteinuria; glomerular disease; hereditary nephropathy; nephropathy
MeSH Terms: conditions — Nephritis, Hereditary; Proteinuria; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective cross-sectional, observational, single-center study of Alport patients, in which a single, first morning voided urine collection will be acquired and used to validate assays of urine biomarkers that reflect changes in glomerular protein filtration barrier function.

The purpose of this study is to identify biomarkers indicative of changes in glomerular filtration function that occur during the course of proteinuric renal diseases such as Alport nephropathy.

ELIGIBILITY:
Inclusion criteria:

* Alport syndrome diagnosis (clinical and/or histopathologic and/or genetic diagnosis, per subject's physician and/or genotyping)
* Physically able to provide a single first-morning urine sample of at least 30 mL

Exclusion criteria:

* Diagnosis of chronic kidney disease
* Receiving chronic phosphate-lowering therapy or erythropoietin therapy
* Ongoing chronic hemodialysis therapy and/or renal transplant recipient
* Nephrotic-range proteinuria: spot urine protein-to-creatinine ratio ≥ 3 on at least 2 of the last 3 clinical assessments Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Alport syndrome identified by the Alport Syndrome Treatments and Outcome Registry (ASTOR)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)